CLINICAL TRIAL: NCT01684072
Title: Evaluation of Safety and Immunogenicity Receiving Live Attenuated Vaccine Against Varicella Without Gelatin
Brief Title: Safety and Immunogenicity Study of Live Attenuated Vaccine Against Varicella Without Gelatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BJCDPC-2
Record Dates: First submitted 2012-09-09; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Chickenpox; Zoster
Keywords: varicella vaccine; gelatin
MeSH Terms: conditions — Chickenpox; Herpes Zoster | interventions — Vaccines; Gelatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vaccine without gelatin (Experimental): use the upper arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: vaccine without gelatin; Biological: vaccine with gelatin
- vaccine with gelatin (Active Comparator): use the upper arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
  Interventions: Biological: vaccine without gelatin; Biological: vaccine with gelatin

INTERVENTIONS:
Biological: vaccine without gelatin — use the upper arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection
Biological: vaccine with gelatin — use the upper arm flank deltoid muscle adheres to stick cohere place the skin after 75% ethyl alcohol disinfection the hypodermic injection

SUMMARY:
The purpose of this study is to observe the occurrence of adverse reaction and antibody positive rate, the elevated level of antibody，Geometric mean titer (GMT) between groups of live attenuated varicella vaccine without gelatin.

DETAILED DESCRIPTION:
Observational Objectives:

To describe the safety of evaluated vaccine, in children aged ≥ 1th birthday and ≤ 12th birthday.

To describe the immunogenicity of evaluated vaccine, in children aged ≥ 1th birthday and ≤ 12th birthday.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent
* Participant is considered to be in good health including the body and mental status on the basis of reported medical history and limited physical examination and live in local ≥ 12 months
* Participant is aged ≥ 1 year to ≤ 12 years
* Body temperature ≤ 37.0℃
* Participant without preventive inoculation of varicella vaccine and previous history of chickenpox and zoster

Exclusion Criteria:

* Known allergy to any constituent of the vaccine
* Reported the history of allergies, convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction
* Known bleeding disorder
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Participation in any other interventional clinical trial
* An acute illness with or without fever (temperature > 37.0℃) in the latest week preceding enrollment in the trial
* Inoculated other vaccines, immunoglobulin or investigational drugs within 4 weeks prior to participation in the study
* Reported clearly the infection of the upper respiratory tract with 6 months
* Clinical Manifestation of Metabolic, blood system, lungs, heart, the gastrointestinal tract, nervous system, kidneys, urinary system, endocrine, liver disease or malignant tumor
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of evaluated vaccine | 8 months
  The immunologic equivalence of 4weeks after vaccination of influenza virus vaccine was measured in terms of the level of antibody.

SECONDARY OUTCOMES:
To evaluate the safety of live attenuated varicella vaccine | 4 months
  The incidence of adverse events was analyzed statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Study Chair — Beijing Chaoyang District Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Chaoyang District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Sanhe Center for Disease Control and Prevention, Langfang, Hebei
  - Jiuyuan Center for Disease Control and Prevention, Baotou, Inner Mongolia